CLINICAL TRIAL: NCT00567177
Title: Objective Measurements of Prolonged Effects of Restasis on Dry Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Richard Yee, MD, Hermann Eye Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-07-0421
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Treatment of Dry Eye Disease
MeSH Terms: interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Restasis, Refresh Plus
- 2 (Placebo Comparator)
  Interventions: Drug: Restasis, Refresh Plus

INTERVENTIONS:
Drug: Restasis, Refresh Plus — Restasis 0.4ml- (in the eye) Instill one drop twice daily in morning and evening Refresh Plus 0.4ml- (in the eye) Instill one drop twice daily in morning and evening

SUMMARY:
We propose to investigate the response to Restasis, over a prolonged period of time in heavy computer users with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Using computers more than three hours per day
* Having dry eye symptoms based on results on the OSDI Scores of 15 or greater on the OSDI will be considered to have the disorder
* An abnormal confocal image of 5 or greater.

Exclusion Criteria:

* All corneal disorders except for tear disorders.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-11; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Dry Eye disease | 6 months

SECONDARY OUTCOMES:
efficacy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Yee, MD, Principal Investigator — Hermann Eye Center
Locations (1):
- Hermann Eye Center, 6400 Fannin Ste 1800, Texas, United States